CLINICAL TRIAL: NCT01608724
Title: A Multicenter, Single Arm, Cohort Study to Evaluate the Efficacy and Safety of Saxagliptin 5mg, Once Daily for 24 Weeks, in Patients With Type 2 Diabetes Mellitus
Brief Title: The Efficacy and Safety Study in Patients With Type 2 Diabetes Mellitus
Acronym: SUNSHINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1680L00008
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental): Saxagliptin, oral 5mg once a day(Q. D.)
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — oral, 5 mg once a day (Q.D.)
  Other Names: Onglyza

SUMMARY:
The efficacy and safety study of saxagliptin 5mg, once daily for 24 weeks in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
A multicenter, single arm, cohort study to evaluate the Efficacy and Safety of saxagliptin 5mg, once daily for 24 weeks, in patients with type 2 diabetes mellitus who are treatment naive or who have inadequate glycaemic control on metformin alone

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures Diagnosed with type 2 diabetes
* Men or women who are >18 years of age at time of consenting upon Visit 1
* HbA1c >7.5% and ≤11.0% Patients should be drug naive or treated with metformin alone on stable doses of for at least continues 8 weeks prior to Visit 1
* Drug naive patients are defined as patients who have not received medical treatment for diabetes (insulin and/or oral hypo)

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Insulin therapy within one year of enrolment (with the exception of insulin therapy during a hospitalization or use in gestational diabetes)
* Previous treatment with any DPP-IV inhibitors or GLP-1 analogue
* History of administration of any antihyperglycemic therapy (other than metformin) during the 8 weeks prior to Visit 1(12 weeks for previous TZD)
* Treatment with systemic glucocorticoids other than replacement therapy
* Inhaled, local injected and topical use of glucocorticoids is allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2165 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Fisher, Study Director — AstraZeneca
Locations (37):
- China (37):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Benxi
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Dongguan
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hhht
  - Research Site, Hubei
  - Research Site, Jimo
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Linyi
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Shiyan
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 92 study centers in China. First subject enrolled: 28 Nov 2012; Last subject last visit: 16 May 2014.
Pre-assignment Details: A total of 2165 patients were screened and 741 patients were excluded due to violation of any inclusion and exclusion criteria.
Groups:
- Saxagliptin: Saxagliptin oral 5mg once a day(Q. D.) for 24 weeks
Period: Overall Study
Arm/Group | Saxagliptin
Started | 1423 (One patient was excluded because the Informed Consent Form was destroyed by site staff by mistake.)
Treated | 1361
Completed | 1180
Not Completed | 243
Not completed — Withdrawal by Subject | 131
Not completed — Lost to Follow-up | 41
Not completed — Study-specific discontinuation criteria | 32
Not completed — Adverse Event | 29
Not completed — Protocol Violation | 6
Not completed — bood sugar too high, etc. | 3
Not completed — Safety reasons | 1

BASELINE CHARACTERISTICS:
Population: Per-protocoal analysis set (PPS), including patients who took at least 1 dose of study drug, had baseline and post-baseline efficacy records, and had no major protocol deviations.
Arm/Group | Saxagliptin
Number analyzed (Participants) | 1210
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.99)
Age, Customized [Number; unit: Participants]
  <65 years | 1063
  >=65 years | 147
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 461
  Male | 749
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1210
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 1210
Baseline haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: %] | 8.85 (0.929)
Baseline fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.08 (2.244)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Haemoglobin A1c (HbA1c)
Description: Evaluation after 24 weeks oral administration of saxagliptin treatment in patients with type 2 diabetes inadequately controlled with diet and exercise or with metformin in addition to diet and exercise.
Time Frame: Weeks 6, 12, and 24
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: (%)
Arm/Group | Saxagliptin
Number analyzed (Participants) | 1210
(%)
  Week 6 | -1.19 (0.033)
  Week 12 | -1.59 (0.039)
  Week 24 | -1.61 (0.040)

2. Secondary Outcome: Proportion (%) of Patients Achieving HbA1c <7%
Time Frame: Weeks 6, 12, and 24
Population: as for baseline characteristics
Measure: Number; unit: Percentage
Arm/Group | Saxagliptin
Number analyzed (Participants) | 1210
Percentage
  Week 6 | 25.4
  Week 12 | 45.6
  Week 24 | 44.1

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Time Frame: Weeks 6, 12, 18, and 24
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin
Number analyzed (Participants) | 1210
mmol/L
  Week 6 | -0.77 (0.063)
  Week 12 | -0.89 (0.065)
  Week 18 | -0.74 (0.071)
  Week 24 | -0.55 (0.070)

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose (2h-PPG)
Time Frame: Week 24
Population: Patients who participated in standard noodle test in the per-protocoal analysis set (PPS), which included patients who took at least 1 dose of study drug, had baseline and post-baseline efficacy records, and had no major protocol deviations.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin
Number analyzed (Participants) | 202
mmol/L | -2.83 (0.274)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Saxagliptin
Serious Adverse Events (participants affected / at risk) | 24/1361
Other Adverse Events (participants affected / at risk) | 69/1361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin (N=1361)
Coronary artery disease (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Diabetic foot infection (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Abortion induced (Surgical and medical procedures) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin (N=1361)
Upper respiratory tract infection (Infections and infestations) | 37
Dizziness (Nervous system disorders) | 36

LIMITATIONS AND CAVEATS:
This was a single-arm study and thus potential placebo effect was unable to be adjusted in any efficacy analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less